CLINICAL TRIAL: NCT06061978
Title: Benefit of Permanent Stimulation of the Left Branch of the His Bundle Versus Right Ventricular Stimulation After Atrioventricular Node Ablation for Rapid Atrial Fibrillation
Acronym: LEANA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/0379/HP
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation Rapid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left bundle branch of His pacing (LBTP) then right ventricular pacing (RVP) (Experimental)
  Interventions: Procedure: left bundle branch of His pacing; Procedure: right ventricular pacing
- right ventricular pacing (RVP) then left bundle branch of His pacing (LBTP) (Experimental)

INTERVENTIONS:
Procedure: left bundle branch of His pacing — left bundle branch of His pacing
  Arms: left bundle branch of His pacing (LBTP) then right ventricular pacing (RVP)
Procedure: right ventricular pacing — right ventricular pacing
  Arms: left bundle branch of His pacing (LBTP) then right ventricular pacing (RVP)

SUMMARY:
The objective of the study is to evaluate the functional benefit of left bundle branch of His pacing compared to right ventricular pacing in patients implanted with a pacemaker prior to a atrioventricular node ablation procedure for rapid atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

1/ Pacemaker implanted patient with LBTP lead and back-up right ventricular lead who subsequently underwent successful atrioventricular node ablation for rapid AF 2) NAV ablation procedure performed less than 15 days ago 3) Age ≥ 18 years 4) Woman of childbearing age with effective contraception (estrogen-progestin or intrauterine device or tubal ligation) for at least 1 month and for the duration of the study, and a negative urine pregnancy test by B-HCG at inclusion Or, Postmenopausal woman: confirmatory diagnosis (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit).

5) Membership of a social security scheme 6) Patient follow-up feasible 7) Patient has read and understood the information leaflet and signed the informed consent form

Exclusion Criteria:

1. Impairment of autonomy such that a maximal cardiorespiratory effort test (VO2 Max test) cannot be performed under good conditions (ADL scale < 5).
2. LVEF < 40% at inclusion
3. Person deprived of liberty by an administrative or judicial decision, or person under court protection, sub-guardianship or curatorship.
4. Patient participating in another interventional trial
5. Any history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol, or from giving informed consent.
6. Pregnant, parturient or breast-feeding women, or those without proven contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Maximum Oxygen Consumption (VO2 max) in mL/min/kg. | 18 months

SECONDARY OUTCOMES:
walking test distance covered | 18 months
echography criteria: LVEF (%), indexed left ventricular end-systolic volume (mL/m2), indexed cardiac output (L/min/m2), inter-ventricular asynchrony criteria (aortic pre-ejection time - pulmonary pre-ejection time) | 18 months
Determination of NT pro BNP or BNP | 18 months
Physical component of quality-of-life scale (SF-36) | 18 months
Medico-economic criteria: incremental cost-utility ratio of LBTP versus RVP | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Corentin CHAUMONT, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de CAEN, Caen, France

IPD SHARING:
Plan to Share IPD: No